CLINICAL TRIAL: NCT04349176
Title: OnabotulinumtoxinA for Chronic Headaches: Is 155 Units Superior to 100 Units?
Brief Title: Onabotulinum Dose Comparison in Chronic Migraine Superior to 100 Units?
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient Recruitment
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sarah Hodges, DO, Principle Investigator, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.2016.0039
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Chronic Migraine, Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A 100U (Experimental)
  Interventions: Drug: Dose
- Group A 155U (Experimental)
  Interventions: Drug: Dose
- Group B 100U (Experimental)
  Interventions: Drug: Dose
- Group B 155 (Experimental)
  Interventions: Drug: Dose

INTERVENTIONS:
Drug: Dose — Randomized to either 100U or 155U

SUMMARY:
The study will enroll patients through the Neurology Department at Naval Medical Center San Diego (NMCSD). Eligible participants will meet criteria for chronic migraine, but will not be excluded based on the presence of significant comorbidities. Participants with comorbidities and medication regimens commonly exhibited within real-world DOD medical settings will not be excluded, such as pain disorders, psychiatric illness, medication overuse, and those who have used prophylactic medication during the baseline period.

This will comprise "Group A". A carefully screened group will comprise "Group B" and meet exclusion criteria designed to approximate that of the PREEMPT2 trial. Within each group, half of the patients (155U Arm) will be randomly selected to receive the standard 155U over 31 fixed sites every 12 weeks while the other half (100U Arm) will receive 100U over 19 fixed sites every 12 weeks. Minimum sample size for the entire cohort is 132 participants (maximum n = 180), with a minimum of 66 participants per comparison.

ELIGIBILITY:
Inclusion Criteria:

Chronic migraine headache - Diagnostic criteria:

A. Headache (tension-type-like and/or migraine-like) on 15 days per month for >3 months2 and fulfilling criteria B and C B. Occurring in a patient who has had at least five attacks fulfilling criteria B-D for 1.1 Migraine without aura and/or criteria B and C for 1.2 Migraine with aura

C. On 8 days per month for >3 months, fulfilling any of the following 3 :

1. criteria C and D for 1.1 Migraine without aura
2. criteria B and C for 1.2 Migraine with aura
3. believed by the patient to be migraine at onset and relieved by a triptan or ergot derivative D. Not better accounted for by another ICHD-3 diagnosis. -

Exclusion Criteria:

Previous exposure at any time to any botulinum toxin serotype Pregnancy, breastfeeding or plans to become pregnant within 6 months Age <18 years Failure to complete at least 20 days of headache diary in the 28 day baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
mean change in frequency of headache days for the baseline period compared to the 28-day period ending with week 24 | 24 weeks

SECONDARY OUTCOMES:
frequency of migraine days | 24 weeks
proportion of patients with severe (>=60) HIT-6 score | 24 weeks
acute headache pain medication intakes | 24 weeks
mean change in total HIT-6 | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No